CLINICAL TRIAL: NCT04533750
Title: Phase I Trial With Expansion Cohort of DNA-PK Inhibition and IMRT in Cisplatin-Ineligible Patients With Stage 3-4 Local-Regionally Advanced Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Testing the Addition of M3814 (Peposertib) to Radiation Therapy for Patients With Advanced Head and Neck Cancer Who Cannot Take Cisplatin
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-06481; NCI-2020-06481 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-HN008 (Other: NRG Oncology); NRG-HN008 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2020-08-29; First posted 2020-09-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Advanced Head and Neck Squamous Cell Carcinoma; Advanced Hypopharyngeal Squamous Cell Carcinoma; Advanced Laryngeal Squamous Cell Carcinoma; Advanced Oral Cavity Squamous Cell Carcinoma; Advanced Oropharyngeal Squamous Cell Carcinoma; Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Stage III Hypopharyngeal Carcinoma AJCC v8; Stage III Laryngeal Cancer AJCC v8; Stage III Lip and Oral Cavity Cancer AJCC v8; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVA Hypopharyngeal Carcinoma AJCC v8; Stage IVA Laryngeal Cancer AJCC v8; Stage IVA Lip and Oral Cavity Cancer AJCC v8; Stage IVA Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVB Hypopharyngeal Carcinoma AJCC v8; Stage IVB Laryngeal Cancer AJCC v8; Stage IVB Lip and Oral Cavity Cancer AJCC v8; Stage IVB Oropharyngeal (p16-Negative) Carcinoma AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Carcinoma | interventions — Fluorodeoxyglucose F18; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy; peposertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (peposertib, IMRT) (Experimental): Beginning 60-90 minutes before each radiation treatment, patients receive peposertib PO QD and undergo IMRT daily Monday-Friday for 7 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, MRI, or 18F-FDG PET/CT during screening and follow-up.
  Interventions: Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Drug: Peposertib; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Other: Fludeoxyglucose F-18 — Given IV
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Peposertib — Given PO
  Other Names: 3-Pyridazinemethanol, alpha-(2-Chloro-4-fluoro-5-(7-(4-morpholinyl)-4-quinazolinyl)phenyl)-6-methoxy-, (alphaS)-; M 3814; M-3814; M3814; MSC 2490484A; MSC-2490484A; MSC2490484A; Nedisertib
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase I trial investigates the side effects and best dose of peposertib when given together with radiation therapy in treating patients with head and neck cancer that has spread to other places in the body (advanced) who cannot take cisplatin. Peposertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. This trial aims to see whether adding peposertib to radiation therapy is safe and works well in treating patients with head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the recommended phase 2 dose (RP2D) of M3814 (peposertib) when given in combination with intensity-modulated radiation therapy (IMRT).

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of the combination of M3814 (peposertib) with radiotherapy.

II. To estimate the rates of grade 3 or greater acute toxicities of the regimen.

III. To estimate late toxicities of the regimen. IV. To evaluate the clinical response rate, based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, at 3 months post completion of radiotherapy.

V. To estimate 6 and 12-month progression-free survival (PFS) in the dose expansion cohort (DEC).

VI. To estimate 6 and 12-month overall survival (OS) in the DEC.

EXPLORATORY OBJECTIVE:

I. To estimate the pharmacokinetic (PK) parameter of M3814 (peposertib) using population PK approaches.

OUTLINE: This is a dose-escalation study of peposertib.

Beginning 60-90 minutes before each radiation treatment, patients receive peposertib orally (PO) once daily (QD) and undergo IMRT daily Monday-Friday for 7 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT), magnetic resonance imaging (MRI), or receive fludeoxyglucose F-18 (18F-FDG) intravenously (IV) and undergo positron emission tomography (PET)/CT during screening and follow-up.

After completion of treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically) proven diagnosis of HNSCC of the oral cavity, oropharynx, larynx, or hypopharynx prior to registration;

  * Patients with oropharynx cancer need p16 determination by immunohistochemistry (where positive is defined as greater than 70% strong nuclear or nuclear and cytoplasmic staining of tumor cells), Note: Institutions must screen patients using a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory. A rigorous laboratory accreditation process similar to the United States (U.S.) CLIA certification, such as the provincial accreditation status offered by the Ontario Laboratory Accreditation (OLA) Program in Canada, the College of American Pathologists (CAP), or an equivalent accreditation in other countries, is acceptable. The p16 results must be reported on the pathology report being submitted;
  * Oral cavity, larynx, hypopharynx, or p16-negative oropharynx cancer must be stages T1-2N2-3 or T3N1-3 or T4N0-3 (American Joint Committee on Cancer [AJCC] version 8);
  * p16-positive oropharynx cancer patients, stages T4N0-3 or T1-3N2-3 (AJCC version 8);
  * The patient has measurable disease as defined by the presence of at least one measurable lesion per RECIST 1.1;
  * Please note: A histological or pathological specimen from cervical lymph nodes with well-defined primary site documented clinically or radiologically is acceptable
* Clinical stage noted above should be based upon following diagnostic workup:

  * History/physical examination within 30 days prior to registration;
  * Examination by radiation oncologist or medical oncologist or otolaryngology (ENT) or head & neck surgeon 30 days prior to registration, including fiber optic exam with laryngopharyngoscopy;
  * Diagnostic quality computed tomography (CT) or magnetic resonance imaging (MRI) of neck, with contrast, within 30 days prior to registration. Fludeoxyglucose F-18 (18F-FDG) whole body positron emission tomography (PET)-CT scan within 42 days of registration is strongly recommended but does not replace the CT or MRI study. Note: If CT component of the PET/CT is of diagnostic quality then PET/CT can be used for eligibility, however the PET/CT scan must be done within 30 days prior to registration
  * Diagnostic quality, cross sectional imaging of the thorax within 42 days prior to registration; 18-F-FDG-PET/CT or conventional CT are acceptable
* Age >= 18 years
* Patients must have a contraindication to cisplatin as defined in the following bullet points. Sites must complete the online tool at comogram.org prior to registration to determine if the patient is eligible. The scores must be recorded on a case report form (CRF). (Refer to data submission table on the NRG-HN008 protocol page on the NRG website);

  * Age >= 70 with moderate to severe comorbidity, defined as having one or more of the following conditions within 30 days prior to registration;

    * Modified Charlson Comorbidity Index >= 1
    * Adult Comorbidity Evaluation (ACE)-27 Index >= 1
    * Omega score < 0.80
    * G-8 score =< 14
    * Cancer and Aging Research Group (CARG) Toxicity Score >= 30%
    * Cumulative Illness Rating Scale for Geriatrics (CIRS-G) Score >= 4 OR
  * Age < 70 with severe comorbidity, defined as having two or more of the following conditions within 30 days prior to registration;

    * Modified Charlson Comorbidity Index >= 1
    * ACE-27 Index >= 1
    * Omega score < 0.80
    * G-8 score =< 14
    * CARG Toxicity Score >= 30%
    * CIRS-G Score >= 4 OR
  * Age >= 18 with an absolute or relative contraindication to cisplatin, defined as one or more of the following criterion within 30 days prior to registration:

    * Pre-existing peripheral neuropathy grade >= 1;
    * Creatinine clearance (CrCl) must be > 30 and < 60 mL/min

      * For this calculation, use the Cockcroft-Gault formula
    * History of hearing loss, defined as either:

      * Existing need of a hearing aid OR
      * >= 25 decibel shift over 2 contiguous frequencies on a pretreatment hearing test as clinically indicated
* Zubrod Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 within 30 days prior to registration
* Whole blood cell (WBC) >= 2000 cells/mm^3 (within 30 days prior to registration)
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3 (within 30 days prior to registration)
* Platelets >= 100,000 cells/mm^3 (within 30 days prior to registration)
* Hemoglobin >= 9.0 g/dL (within 30 days prior to registration); Note: The use of transfusion is acceptable
* Creatinine clearance (CrCl) > 30 mL/min (within 30 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (except patients with Gilbert syndrome who can have total bilirubin < 3.0 mg/dL) (within 30 days prior to registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN (within 30 days prior to registration)
* For women of child bearing potential (e.g. uterus present and menstruating), a negative serum pregnancy test within 14 days prior to registration. Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL
* The patient must provide study-specific informed consent prior to study entry
* Known human immunodeficiency virus (HIV) infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months and CD4 T cell count >= 200 are eligible for this trial. Testing is not required for entry into protocol
* Patients with a history of hepatitis B or C infection are eligible if they have an undetectable viral load
* Willing to use highly effective contraceptives for males and females of childbearing potential during therapy and for 12 weeks after the last dose of M3814 (peposertib); this inclusion is necessary because the treatment in this study may be significantly teratogenic
* Patients must be able to swallow whole tablets

Exclusion Criteria:

* Definitive clinical or radiologic evidence of distant (beyond cervical lymph node and neck tissue) metastatic disease
* Carcinoma of the neck of unknown primary site origin
* Patients with oral cavity cancer are excluded from participation if the patient is medically operable and the resection of the primary tumor is considered technically feasible by an oral or head and neck cancer surgical subspecialist
* Gross total excision of both primary and nodal disease; this includes tonsillectomy, local excision of primary site, and nodal excision that removes all clinically and radiographically evident disease

  * Note: Patients with RECIST, version (v.) 1.1 evaluable remaining cancer either in the neck or primary site remain eligible
* Prior invasive malignancy (except non-melanomatous skin cancer carcinoma, in situ of the breast, oral cavity, or cervix, low or very low-risk prostate cancer) unless disease free for a minimum of 3 years
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable if not within =< 3 years
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Severe, active co-morbidity defined as follows:

  * History of bone marrow transplant and organ transplant, including allogenic stem cell transplantation;
  * Unstable angina requiring hospitalization in the last 6 months;
  * New York Heart Association Functional classification III/IV (Note: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification.);
  * Myocardial infarction within the last 6 months;
  * Persistent grade 3-4 (Common Terminology Criteria for Adverse Events [CTCAE] version 5.0) electrolyte abnormalities that cannot be reversed despite as indicated by repeat testing;
  * Ongoing active infection that is associated with symptoms and/or requires antibiotic therapy at the time of registration (excluding asymptomatic bacteriuria, genital herpes, oral herpes, thrush, bacterial vaginosis, vaginal candidiasis, topical antifungals)
* Pregnancy and nursing females, if applicable
* Concomitant use of proton pump inhibitors (or unable to stop 5 days prior to treatment)
* Receipt of live vaccinations within 28 days prior to registration
* Patients unable to discontinue medications or substances that are:

  * Strong inhibitors, inducers or sensitive substrates of CYP3A4/5, CYP2C19, or CYP2C9 prior to study treatment;
  * Substrates of CYP1A2, CYP2B6, or CYP3A4/5 with a narrow therapeutic prior to study treatment;

    * Note: Opioids are allowed, with the exception of methadone
* Fridericia's correction formula (QTcF) > 450 ms for males and > 470 ms for females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2025-12-07 (Actual); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Up to 28 days after the end of intensity-modulated radiation therapy (IMRT)

SECONDARY OUTCOMES:
Incidence of acute toxicity | Up to 3 months from IMRT completion
  Will be as measured by Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0
Incidence of late toxicity | More than 3 months from IMRT completion for up to 2 years
  Will be as measured by CTCAE v5.0.
Clinical response rate | At 3 months post completion of IMRT
  Will be assessed by Response Evaluation Criteria in Solid Tumors 1.1.
Progression-free survival (PFS) rates | At 6 months and 1 year
  Will be estimated using the Kaplan-Meier (K-M) method (Kaplan and Meier 1958). Point estimates of the PFS at 6 months and 1 year post-IMRT along with their 95% confidence intervals after using a log-log transformation will be calculated using the K-M curves.
Overall survival (OS) rates | At 6 months and 1 year
  Will be estimated using the Kaplan-Meier (K-M) method (Kaplan and Meier 1958). Point estimates of the OS at 6 months and 1 year post-IMRT along with their 95% confidence intervals after using a log-log transformation will be calculated using the K-M curves.

OTHER OUTCOMES:
Pharmacokinetic (PK) parameter of M3814 (peposertib) | Within 30 minutes before administration, 2 hours and 4 hours after administration on day 1 of weeks 1 and 2
  Plasma PK values will be estimated in the context of the Merck popPK model at the end of the trial and reported as such. PK-outcome relationships may be assessed in an exploratory fashion.

CONTACTS AND LOCATIONS:
Overall Officials: Maura L Gillison, Principal Investigator — NRG Oncology
Locations (27):
- United States (27):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - M D Anderson Cancer Center, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2024-08-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT04533750/ICF_000.pdf